CLINICAL TRIAL: NCT03645928
Title: A Phase 2, Multicenter Study of Autologous Tumor Infiltrating Lymphocytes (LN 144/LN-145/LN-145-S1) in Patients With Solid Tumors
Brief Title: Study of Autologous Tumor Infiltrating Lymphocytes in Patients With Solid Tumors
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Iovance Biotherapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IOV-COM-202; 2018-001608-12 (EudraCT Number); 2024-510779-39-00 (EU CTIS Number)
Record Dates: First submitted 2018-08-22; First posted 2018-08-24 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Metastatic Melanoma; Squamous Cell Carcinoma of the Head and Neck; Non-small Cell Lung Cancer
Keywords: LN-144; LN-145; Cell Therapy; Autologous Adoptive Cell Transfer; Autologous Adoptive Cell Therapy; Cellular Immuno-therapy; Tumor Infiltrating Lymphocytes; TIL; IL-2; Multiple Tumor Type; Lifileucel; Pembrolizumab; LN-145-S1; Ipilimumab; Nivolumab; ICI; Immune Checkpoint Inhibitor; Aldesleukin; Nivolumab-relatlimab; Platinum doublet chemotherapy agents; Cisplatin; Carboplatin; Paclitaxel; Nab-Paclitaxel; Non-small cell lung cancer; Melanoma
MeSH Terms: conditions — Melanoma; Squamous Cell Carcinoma of Head and Neck; Carcinoma, Non-Small-Cell Lung | interventions — lifileucel; Toll-Like Receptor 1; pembrolizumab; Ipilimumab; Nivolumab; Opdualag; Cisplatin; Carboplatin; Paclitaxel; 130-nm albumin-bound paclitaxel; Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (10):
- Cohort 1A (Experimental): LN-144 therapy in combination with pembrolizumab in patients with Stage IIIC to IV unresectable or metastatic melanoma with ≤ 3 prior lines of systemic therapy, excluding immune checkpoint inhibitors (ICI).
  Interventions: Biological: Lifileucel; Drug: Pembrolizumab
- Cohort 1B (Experimental): LN-145-S1 therapy as a single agent in patients with Stage IIIC or Stage IV unresectable or metastatic melanoma, who have previously received systemic therapy with a PD-1 blocking antibody. If the tumor is proto-oncogene B-Raf (BRAF) V600 mutation positive, patients must have received a BRAF inhibitor with or without a mitogen-activated extracellular signal-related kinase (MEK) inhibitor.
  Interventions: Biological: LN-145-S1
- Cohort 1C (Experimental): LN-144 Generation 3 (Gen 3) therapy as a single agent in patients with Stage IIIC or Stage IV unresectable or metastatic melanoma, who have previously received systemic therapy with a PD-1 blocking antibody. If the tumor is BRAF V600 mutation positive, patients must have received BRAF inhibitor with or without a MEK inhibitor.
  Interventions: Biological: Lifileucel
- Cohort 2A (Experimental): LN-145 therapy in combination with pembrolizumab in patients with advanced, recurrent, or metastatic HNSCC, with ≤ 3 prior lines of systemic therapy, excluding ICIs.
  Interventions: Biological: LN-145; Drug: Pembrolizumab
- Cohort 3A (Experimental): LN-145 therapy in combination with pembrolizumab in patients with locally advanced or metastatic (Stage III or Stage IV) non-small-cell lung cancer (NSCLC) with ≤ 3 prior lines of systemic therapy, excluding ICIs, or ≤ 4 lines if 2 or more of the lines are TKI therapy for those with tumors that harbored actionable mutations (eg, EGFR, ALK, ROS).
  Interventions: Biological: LN-145; Drug: Pembrolizumab
- Cohort 3B (Experimental): LN-145 therapy as a single agent in patients with Stage III or Stage IV NSCLC, who have previously received 1-3 lines of prior systemic therapy. Patients with known oncogene drivers (eg, EGFR, ALK, ROS) who have mutations that are sensitive to targeted therapies are not required to have received prior systemic therapy with ICIs.
  Interventions: Biological: LN-145
- Cohort 3C (Experimental): LN-145 therapy in combination with ipilimumab and nivolumab in patients with Stage III or Stage IV NSCLC who have previously received 1 line of ICI monotherapy. No other systemic therapy for metastatic disease is allowed. Prior chemoradiation and/or chemotherapy in the adjuvant and/or neo-adjuvant settings are allowed.
  Interventions: Biological: LN-145; Drug: Ipilimumab; Drug: Nivolumab
- Cohort 1D (Experimental): The lifileucel regimen in combination with nivolumab-relatlimab in patients with Stage IIIC to IV unresectable or metastatic (advanced) melanoma who have had no prior therapy for advanced disease.
  Interventions: Biological: Lifileucel; Drug: Nivolumab-relatlimab
- Cohort 3D (Experimental): The lifileucel regimen in combination with pembrolizumab with or without pemetrexed, after tumor resection before 4 cycles of frontline platinum doublet chemotherapy plus pembrolizumab, in patients with Stage IV NSCLC without EGFR, ALK, or ROS1 driver mutations, who have had no prior therapy for advanced disease.
  Interventions: Biological: Lifileucel; Drug: Pembrolizumab; Drug: Cisplatin; Drug: Carboplatin; Drug: Paclitaxel; Drug: Nab-Paclitaxel; Drug: Pemetrexed
- Cohort 3E (Experimental): The lifileucel regimen in combination with pembrolizumab with or without pemetrexed, after tumor resection during 4 cycles of frontline platinum doublet chemotherapy plus pembrolizumab, in patients with Stage IV NSCLC without EGFR, ALK, or ROS1 driver mutations.
  Interventions: Biological: Lifileucel; Drug: Pembrolizumab; Drug: Cisplatin; Drug: Carboplatin; Drug: Paclitaxel; Drug: Nab-Paclitaxel; Drug: Pemetrexed

INTERVENTIONS:
Biological: Lifileucel — A tumor sample is resected from each patient and cultured ex vivo to expand the population of tumor infiltrating lymphocytes. After NMA lymphodepletion, patients are infused with Lifileucel followed by aldesleukin administration. Lifileucel will be administered to patients once (on Day 0) during the study.
  Other Names: LN-144/LN-145, TIL, autologous tumor infiltrating lymphocytes, lifileucel
  Arms: Cohort 1A; Cohort 1C; Cohort 1D; Cohort 3D; Cohort 3E
Biological: LN-145 — A tumor sample is resected from each patient and cultured ex vivo to expand the population of tumor infiltrating lymphocytes. After NMA lymphodepletion, patients are infused with their autologous TIL (LN-145) followed by aldesleukin administration. TIL will be administered to patients once (on Day 0) during the study.
  Other Names: TIL, autologous tumor infiltrating lymphocytes
  Arms: Cohort 2A; Cohort 3A; Cohort 3B; Cohort 3C
Drug: Pembrolizumab — Humanized antibody.
  Pembrolizumab will be administered following tumor resection and will continue every 3 weeks or every 6 weeks thereafter for up to 2 years.
  Other Names: Keytruda
  Arms: Cohort 1A; Cohort 2A; Cohort 3A; Cohort 3D; Cohort 3E
Biological: LN-145-S1 — A tumor sample is resected from each patient and cultured ex vivo to expand the population of tumor infiltrating lymphocytes. After NMA lymphodepletion, patients are infused with their autologous TIL (LN-145-S1) followed by aldesleukin administration. TIL will be administered to patients once (on Day 0) during the study.
  Other Names: TIL, autologous tumor infiltrating lymphocytes
  Arms: Cohort 1B
Drug: Ipilimumab — Monoclonal antibody
  Ipilimumab will be administered as a single dose prior to tumor resection.
  Other Names: Yervoy
  Arms: Cohort 3C
Drug: Nivolumab — Monoclonal antibody
  Nivolumab will be administered once prior to tumor resection. The second dose will be administered prior to TIL administration and dosing will continue every 4 weeks for up to 2 years.
  Other Names: Opdivo
  Arms: Cohort 3C
Drug: Nivolumab-relatlimab — Nivolumab-relatlimab will be administered following tumor resection and will continue every 4 weeks thereafter for up to 2 years.
  Other Names: Opdualag
  Arms: Cohort 1D
Drug: Cisplatin — Cisplatin administered intravenously at the protocol-defined dose every 3 weeks for up to 4 cycles.
  Arms: Cohort 3D; Cohort 3E
Drug: Carboplatin — Carboplatin administered intravenously at the protocol-defined dose every 3 weeks for up to 4 cycles.
  Arms: Cohort 3D; Cohort 3E
Drug: Paclitaxel — Paclitaxel administered intravenously at the protocol-defined dose every 3 weeks for up to 4 cycles.
  Arms: Cohort 3D; Cohort 3E
Drug: Nab-Paclitaxel — Nab-Paclitaxel administered intravenously at the protocol-defined dose every 3 weeks for up to 4 cycles.
  Arms: Cohort 3D; Cohort 3E
Drug: Pemetrexed — Pemetrexed administered intravenously at the protocol-defined dose every 3 weeks for up to 4 cycles. Optional continuation maintenance every 3 weeks, if applicable.
  Arms: Cohort 3D; Cohort 3E

SUMMARY:
A prospective, open-label, multi-cohort, non-randomized, multicenter Phase 2 study evaluating adoptive cell therapy (ACT) with TIL [LN-144/LN-145 (lifileucel)] in combination with immune checkpoint inhibitors or TIL [LN-144/LN-145 (lifileucel) and LN-145-S1] as a single agent therapy.

DETAILED DESCRIPTION:
TIL [LN-144/LN-145 (lifileucel) and LN-145-S1] is an adoptive cell transfer therapy that utilizes an autologous TIL for the treatment of patients with unresectable or metastatic melanoma, advanced, recurrent, or metastatic squamous cell carcinoma of the head and neck, and locally advanced or metastatic non-small cell lung cancer. The adoptive cell transfer therapy used in this study involves patients receiving a nonmyeloablative (NMA) lymphodepletion regimen, followed by infusion of autologous TIL followed by the administration of aldesleukin. Patients in Cohorts 1A, 1D, 2A, 3A, 3C, 3D, and 3E will receive TIL plus immune checkpoint inhibitors. Patients in Cohorts 1B, 1C, and 3B will receive autologous TIL as a single therapy.

ELIGIBILITY:
Inclusion Criteria

* Must have a confirmed diagnosis of malignancy of their receptive histologies: unresectable or metastatic melanoma Stage IIIC to IV (Cohorts 1A,1B and 1C), advanced, recurrent or metastatic HNSCC (Cohort 2A), or Stage III or Stage IV non-small cell lung cancer (Cohorts 3A, 3B, and 3C). Stage IV NSCLC with no actionable mutations (EGFR, ALK, ROS1) with effective targeted therapy (Cohorts 3D and 3E).
* Cohorts 1A, 1D, 2A, 3A, 3D and 3E: If previously treated, patients must have progressed on or after most recent therapy and must not have received ICIs as part of one of the counted lines of prior therapy. Patients must have radiologically documented disease progression while receiving or after the completion of the most recent prior treatment. Patients may have received up to 3 prior systemic anticancer therapies (except for Cohort 3A, where patients whose tumors harbor actionable mutations may have received up to 4 prior systemic therapies). Patients in Cohort 1D may have had no prior therapy for advanced disease. Patients in Cohorts 3D and 3E may have had no prior systemic therapy for Stage IV disease.
* Cohorts 1B, 1C, 3B, and 3C: Unresectable or metastatic melanoma patients in Cohorts 1B or 1C must have previously received systemic therapy with a PD-1 blocking antibody. NSCLC patients in Cohort 3B must have previously received systemic therapy with any ICI (except for those patients with known oncogene driver mutations that are sensitive to targeted therapies) as part of 1 - 3 prior lines of therapy. NSCLC patients in Cohort 3C must have previously received 1 line of ICI monotherapy. No other systemic therapy for metastatic disease is allowed. Prior chemoradiation and/or chemotherapy in the adjuvant and/or neoadjuvant settings are allowed.
* Must have at least 1 resectable lesion
* Must have remaining measurable disease as defined by RECIST 1.1 following tumor resection
* Must be ≥ 18 years at the time of consent for Cohorts 1A, 1C, 1D, 2A, 3A, 3B, 3C, 3D and 3E. Patients must be ≥ 12 years at the time of consent for Cohort 1B. Enrollment of patients > 70 years of age may be allowed after consultation with the Medical Monitor.
* Must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1, and an estimated life expectancy of ≥ 6 months.
* Patients of childbearing potential or those with partners of childbearing potential must be willing to practice an approved method of birth control during treatment and for 12 months after their last dose of aldesleukin, 4 months after their last dose of pembrolizumab, 5 months after their last dose of ipilimumab or nivolumab, or nivolumab-relatlimab; 6 months after the last dose of carboplatin; 14 months after the last dose of cisplatin; and 6 months after the last dose of pemetrexed, paclitaxel, or nab-paclitaxel, whichever occurs later.

Exclusion Criteria

* Patients with melanoma of uveal/ocular origin.
* Patients who have a history of allogeneic organ transplant or any form of cell therapy involving prior conditioning chemotherapy within the past 20 years. Patients being retreated with TIL, as part of this study are not excluded.
* Patients who have symptomatic, untreated brain metastases or history of leptomeningeal metastases.
* Patients who are on systemic steroid therapy > 10 mg/day of prednisone or other steroid equivalent. Patients receiving steroids as replacement therapy for adrenocortical insufficiency at ≤ 10 mg/day of prednisone or other steroid equivalent may be eligible.
* Patients who are pregnant or breastfeeding.
* Patients who have an active medical illness(es), which in the opinion of the Investigator, would pose increased risks for study participation
* Cohort 1A, 1D, 2A, 3A, 3C, 3D and 3E patients may not have a medical history of autoimmune disorders (including pneumonitis) requiring treatment or active management.
* Patients who have received a live or attenuated vaccination within 28 days prior to the start of treatment
* Patients who have any form of primary immunodeficiency
* Patients with a history of hypersensitivity to any component of the study drugs to be administered in the pertinent cohort(s).
* Patients who have a left ventricular ejection fraction (LVEF) < 45% or who are New York Heart Association Class II or higher. A cardiac stress test demonstrating any irreversible wall movement abnormality in any patients ≥60 years of age or in patients who have a history of ischemic heart disease, cardiac chest pain, or clinically significant atrial and/or ventricular arrhythmias.
* Patients with respiratory dysfunction or history of smoking are excluded if not meeting either of forced expiratory volume in 1 second (FEV1)/forced vital capacity (FVC) > 0.7 or FEV1 > 50%.
* Patients who have had another primary malignancy within the previous 3 years
* Participation in another interventional clinical study within 21 days prior to the initiation of treatment.
* Patients in Cohorts 1D, 3D, or 3E who previously received adjuvant or neoadjuvant ICI(s) for non-metastatic disease and had an immune-related AE(s) requiring systemic steroid treatment or discontinuation of immune checkpoint inhibitor therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 245 (Estimated)
Dates: Start 2019-05-07 (Actual); Primary Completion 2029-08-09 (Estimated); Study Completion 2029-08-09 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | Up to 60 months
  To evaluate the efficacy of autologous TIL in combination with ICIs in metastatic melanoma, HNSCC, and NSCLC patients and as a single therapy in metastatic melanoma and NSCLC patients as determined by objective response rate (ORR) using the Response Evaluation Criteria in Solid Tumors (RECIST 1.1) as assessed by Investigator
Safety Profile Measured by Grade ≥3 TEAEs | Up to 60 months
  To characterize the safety profile of autologous TIL in combination with ICIs in metastatic melanoma, HNSCC, and NSCLC patients and as a single therapy in metastatic melanoma and NSCLC patients as measured by the incidence of Grade ≥ 3 treatment-emergent adverse events (TEAEs)
To evaluate the feasibility of producing lifileucel using tumor samples obtained before (Cohort 3D) or during (Cohort 3E) frontline platinum doublet chemotherapy and pembrolizumab in patients with Stage IV NSCLC | Up to 60 months
  Feasibility is measured by the percentage of patients for whom lifileucel is successfully manufactured and meets release specification and defined as the number of patients with lifileucel product that meets specification divided by the total number of patients who had tumor resection.

SECONDARY OUTCOMES:
Complete Response Rate | Up to 60 months
  To evaluate efficacy parameters such Complete Response (CR) rate per RECIST 1.1, as assessed by the Investigator
Duration of Response | Up to 60 months
  To evaluate efficacy parameters such Duration of Response (DOR) per RECIST 1.1, as assessed by the Investigator
Disease Control Rate | Up to 60 months
  To evaluate efficacy parameters such Disease Control Rate (DCR) per RECIST 1.1, as assessed by the Investigator
Progression-Free Survival | Up to 60 months
  To evaluate efficacy parameters such Progression-Free Survival (PFS) per RECIST 1.1, as assessed by the Investigator
Overall Survival | Up to 60 months
  To evaluate efficacy parameters such Overall Survival (OS)

CONTACTS AND LOCATIONS:
Overall Officials: Iovance Biotherapeutics Medical Monitor, Study Director — Iovance Biotherapeutics
Locations (45):
- United States (24):
  - University of California, San Diego, La Jolla, California
  - University of Southern California, Los Angeles, California
  - University of California, Los Angeles, Los Angeles, California
  - University of Colorado, Denver, Colorado
  - Yale University, New Haven, Connecticut
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - Mount Sinai Medical Center, Miami Beach, Florida
  - Orlando Health Cancer Institute, Orlando, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - University of Louisville, Louisville, Kentucky
  - University of Maryland, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - MD Anderson at Cooper, Camden, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Columbia University, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of Cincinnati, Cincinnati, Ohio
  - Ohio State University, Columbus, Ohio
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Huntsman Cancer Hospital, Salt Lake City, Utah
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada
- Centre Léon Berard, Lyon, France
- Germany (3):
  - Klinikum rechts der Isar der Technischen Universität München, München, Bavaria
  - Universitätsklinikum Carl Gustav Carus, Dresden, Saxony
  - Universitätsklinikum Schleswig-Holstein - Campus Lübeck, Lübeck, Schleswig-Holstein
- Greece (2):
  - Laiko General Hospital of Athens, Athens, Attica
  - Attikon University General Hospital, Athens, Attica
- Spain (8):
  - Hospital Universitario Marques de Valdecilla, Santander, Cantabria
  - Hospital Regional Universitario de Malaga - Hospital General, Málaga, Málaga
  - University Hospital Vall d'Hebron, Barcelona
  - ICO l'Hospitalet - Hospital Duran i Reynals, Barcelona
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospital Universitario Fundacion Jimenez Diaz, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario HM Sanchinarro, Madrid
- Switzerland (3):
  - Universitätsspital Basel, Basel
  - Universitaetsspital Bern, Bern
  - Centre Hospitalier Universitaire Vaudois, Lausanne
- United Kingdom (3):
  - Guy's Hospital, London, England
  - The Royal Marsden NHS Foundation Trust, London, England
  - Bristol Haematology and Oncology Centre, Bristol

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hensel J, Metts J, Gupta A, Ladle BH, Pilon-Thomas S, Mullinax J. Adoptive Cellular Therapy for Pediatric Solid Tumors: Beyond Chimeric Antigen Receptor-T Cell Therapy. Cancer J. 2022 Jul-Aug 01;28(4):322-327. doi: 10.1097/PPO.0000000000000603. PMID 35880942